CLINICAL TRIAL: NCT02638636
Title: Internet-based Exposure-based Therapy for Fibromyalgia: A Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, Med Dr., Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPN 2015/1528-31/1
Record Dates: First submitted 2015-12-17; First posted 2015-12-23 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Fibromyalgia
Keywords: Cognitive behavior therapy; Randomized controlled trial; Exposure therapy; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based exposure therapy (Experimental): The experimental group will go through active internet-based treatment which is delivered on a safe internet platform. Treatment is divided into eight modules, each containing homework assignments. Participants in experimental group will be assigned a therapist that they can contact through a message system in the platform and expect answer within 48 hours.
  Interventions: Behavioral: Internet-based exposure therapy
- Waitlist (No Intervention): Waitlist control, i.e. no active active intervention during waiting list period. Will be offered treatment when the first group has finished (i.e. week 10).

INTERVENTIONS:
Behavioral: Internet-based exposure therapy — The treatment is a 10 week long cognitive behavior therapy. It is based mainly on the principles of exposure; i.e. the participant is instructed to approach situations they have avoided in order to reduce or avoid pain or other aversive experiences until they feel less discomfort and extended behavior repertoire in presence of pain and aversive inner experiences Other interventions include psychoeducation, mindfulness and acceptance strategies and are employed in order to facilitate exposure.
  Arms: Internet-based exposure therapy

SUMMARY:
The purpose of this study is to examine if an internet-based exposure therapy is effective in reducing Fibromyalgia symptoms and impact amongst patients with Fibromyalgia.

DETAILED DESCRIPTION:
Trial Objectives: Primary objective is to investigate whether an Internet-based exposure therapy can effectively reduce the degree of Fibromyalgia symptoms and impact. Secondary objectives are to 1) investigate the treatment's ability to reduce degree of a) quality of life b) function c) insomnia and fatigue d) pain-related fear and negative thoughts e) depression and anxiety, cost-effectiveness of this treatment; and 2) to study if any variables could moderate/mediate the treatment outcome, such as a) degree of covert avoidance, b) degree of reactivity to inner sensations

Trial Design: Randomized controlled trial with waitlist control, who also will receive treatment after the first group has finished.

Duration: Ten weeks

Primary Endpoint: Change in Fibromyalgia symptoms and impact from baseline to Week 10. Long term follow-up is also investigated (potential changes from post-treatment to 6- and 12 months after treatment completion)

Efficacy Parameters: the Fibromyalgia Impact Questionnaire (FIQ)

Description of Trial Subjects: Patients > 18 years old, Fibromyalgia diagnosis, residing in Sweden.

Number of Subjects: 140

Sample size estimation: Sample size is based on a estimated effect size (measured by Cohen's d) of 0.5, based on a power of 0.8 and with room for a 10 % dropout rate.

Recruitment: Self-referral. Advertising will be made through national newspaper, social media and on patient organisations' websites.

Safety parameters: Participants will have the opportunity to report any adverse events during treatment at posttreatment and follow-up measurements.

Data collection: Data will be collected electronically via the treatment platform.

Plan for missing data: Last-observation carried forward (LOCF).

Main statistical analysis: Hierarchical linear mixed modelling.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia diagnosis
* Swedish resident
* Internet connection before, under and after treatment
* Willing to refrain from other concurrent psychological treatment during the study
* Agreement to keep psychotrophic medication constant during the study

Exclusion Criteria:

* Severe depression (≥30 points on Montgomery Åsberg Depression Rating Scale - Self Rated (MADRS-S) or risk of suicide (≥4 points on the suicide item on MADRS-S)
* Ongoing alcohol or substance abuse
* Psychosis
* Other severe illness that require immediate treatment and/or was considered the participants primary concern other than FM, or bodily condition that makes treatment unfeasible (such as late pregnancy; >29 weeks gestation
* Illiteracy or poor skills in Swedish language
* Insufficient computer or language skills to manage a text-based treatment.
* Other concurrent psychological treatment
* Recent changes in psychotrophic medication (<6 weeks prior to randomization)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in the Fibromyalgia Impact Questionnaire (FIQ) | Week 0, week 10, Long term follow-up at 6- and 12-months after treatment has ended]
  Change in Fibromyalgia symptoms and impact from baseline to Week 10, and at 6- and 12 months after treatment has ended.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Week 0, week 10, follow-up at 6- and 12-months after treatment has ended
  Change in sleep disturbances from baseline to Week 10, and at 6- and 12 months after treatment has ended.
Fatigue Severity Scale (FSS) | Week 0, week 10, follow-up at 6- and 12-months after treatment has ended
  Change in fatigue from baseline to Week 10, and at 6- and 12 months after treatment has ended.
WHO Disability Assessment Schedule 2.0 (WHODAS 2) | Week 0, week 10, follow-up at 6- and 12-months after treatment has ended
  Change in level of function from baseline to Week 10, and at 6- and 12 months after treatment has ended.
Brunnsviken Brief Quality of Life Inventory (BBQ) | Week 0, week 10, follow-up at 6- and 12-months after treatment has ended
  Change in quality of life from baseline to Week 10, and at 6- and 12 months after treatment has ended.
The Psychological Inflexibility in Pain Scale (PIPS) | Week 0, week 10, follow-up at 6- and 12-months after treatment has ended
  Change in covert avoidance from baseline to Week 10, and at 6- and 12 months after treatment has ended.
Pain Reactivity Scale (PRS) | Week 0, week 10, follow-up at 6- and 12-months after treatment has ended
  Change in pain-related fear and negative thoughts from baseline to Week 10, and at 6- and 12 months after treatment has ended.
Patient Health Questionnaire-9 (PHQ-9) | Week 0, week 10, follow-up at 6- and 12-months after treatment has ended
  Change in level of depression from baseline to Week 10, and at 6- and 12 months after treatment has ended.
Generalised Anxiety Disorder 7-item scale (GAD-7) | Week 0, week 10, follow-up at 6- and 12-months after treatment has ended
  Change in level of anxiety from baseline to Week 10, and at 6- and 12 months after treatment has ended.
Subscale "reactivity to inner experiences" from Five Facets of Mindfulness Questionnaire (FFMQ) | Week 0, week 10, follow-up at 6- and 12-months after treatment has ended
  Change in reactivity to inner experiences from baseline to Week 10, and at 6- and 12 months after treatment has ended.
Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) | Week 0, week 10, follow-up at 6- and 12-months after treatment has ended
  Change in health-care costs and sick-leave from baseline to Week 10, and at 6- and 12 months after treatment has ended.
EQ5D | Week 0, week 10, follow-up at 6- and 12-months after treatment has ended
  Change in health-related quality of life from baseline to week 10, and at 6- and 12 months after treatment has ended.

OTHER OUTCOMES:
Item 9 from Montgomery Asberg Depression Rating Scale (MADRS-S) | Week 1, week 2, week 3, week 4, week 5, week 6, week, 7, week 8, week 9
  Possible presence of suicidal thoughts or ideation during treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hedman-Lagerlof M, Andersson E, Ljotsson B, Engelbrektsson J, Lundback K, Bjorkander D, Hedman-Lagerlof E, Flink I, Axelsson E. Effect moderators in Internet-based exposure therapy for fibromyalgia: The role of pain intensity. Eur J Pain. 2023 Apr;27(4):507-517. doi: 10.1002/ejp.2074. Epub 2023 Jan 10. PMID 36585933